CLINICAL TRIAL: NCT04157075
Title: The Effect of Intra-operative Uterosacral Bupivacaine Injection on Post-operative Pain in Patients Undergoing Minimally Invasive Hysterectomy
Brief Title: Intra-operative Uterosacral Ligament Bupivacaine Injection During Minimally Invasive Hysterectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00221267
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-03

CONDITIONS: Pain, Postoperative; Opioid Use
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded to which arm they are in, surgeon will not as they will be performing injection however will not be assessing pain scores
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- No injection (Placebo Comparator): No injection will be performed
  Interventions: Drug: Bupivacaine
- Normal Saline Injection (Sham Comparator): Normal saline will be injected into the uterosacral ligaments prior to colpotomy
  Interventions: Drug: Bupivacaine
- Bupivacaine Injection (Active Comparator): Bupivacaine will be injected into the uterosacral ligaments prior to colpotomy
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Bupivicaine injection into uterosacral ligaments prior to colpotomy

SUMMARY:
This is proof of concept, phase I randomized controlled trial studying a short acting non-opioid anesthetic, bupivacaine to improve post-operative pain in gynecologic surgery patients. Patients who are undergoing minimally invasive (laparoscopic or robotic) hysterectomy will be randomized to receive no uterosacral injection, normal saline uterosacral injection, or 0.25% bupivacaine uterosacral injection just prior to colpotomy (incision around the cervix and removal of uterus) during minimally invasive hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 years old
* undergoing benign minimally invasive hysterectomy with minimally invasive GYN surgeon at Johns Hopkins Hospital
* Patients must be English speaking.

Exclusion Criteria:

* Pregnancy
* allergy, contraindication, or intolerance to bupivacaine, opioids, Tylenol, or NSAID drugs
* pre-operative daily opioid consumption
* peri-operative transverse abdominis plane block
* recent history of drug or alcohol abuse (in last year)
* severe cardiovascular, hepatic or renal disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Difference in post-operative opioid usage with the use of uterosacral ligament bupivacaine injection | 7 days post-op
  Total morphine equivalents of opioids in the first 7 days after surgery will be assessed to look for a statistically significant difference

SECONDARY OUTCOMES:
Difference in Visual analog scores (VAS) scores following uterosacral ligament bupivicaine injection | 7 days post-op
  Patient will report VAS scores daily until post-op day 7 on a scale of 1-10 with higher scores indicating higher pain severity. The investigators will be looking for a statistically significant difference between the treatment and placebo vs. sham group.
Time to first bowel movement following uterosacral ligament bupivicaine injection | 7 days post-op
  Patients will record when they resume normal bowel function on a pill diary post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Karen Wang, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Howard County General Hospital, Columbia, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frost AS, Kohn JR, Le Neveu M, Brah T, Okonkwo O, Borahay MA, Wu H, Simpson K, Patzkowsky KE, Wang KC. Laparoscopic administration of bupivacaine at the uterosacral ligaments during benign laparoscopic and robotic hysterectomy: a randomized controlled trial. Am J Obstet Gynecol. 2023 Nov;229(5):526.e1-526.e14. doi: 10.1016/j.ajog.2023.07.047. Epub 2023 Jul 31. PMID 37531986